CLINICAL TRIAL: NCT02325557
Title: A Phase 1-2 Dose-Escalation and Safety Study of ADXS31-142 Alone and of ADXS31-142 in Combination With Pembrolizumab (MK-3475) in Patients With Previously Treated Metastatic Castration-Resistant Prostate Cancer
Brief Title: ADXS31-142 Alone and in Combination With Pembrolizumab (MK-3475) in Participants With Previously Treated Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADXS142-03; KEYNOTE-046 (Other: Merck)
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Prostate Cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: ADXS31-142 (Experimental): Participants received ADXS31-142 1 × 10^9 colony-forming units (CFU), 5 × 10^9 CFU, or
  1 × 10^10 CFU intravenously (IV) every 3 weeks (Q3W) in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
  Interventions: Drug: ADXS31-142
- Part B: ADXS31-142 + Pembrolizumab (Experimental): Participants received ADXS31-142 1 × 10^9 CFU) IV Q3W (in a 12-week cycle) in combination with 200 mg pembrolizumab IV Q3W for three times, with a fourth pembrolizumab dose 3 weeks later (in 12 week-cycles) for up to 24 months or until disease progression or discontinuation.
  Interventions: Drug: ADXS31-142; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ADXS31-142 — ADXS31-142 IV infusion
Drug: Pembrolizumab — Pembrolizumab IV infusion
  Other Names: MK-3475
  Arms: Part B: ADXS31-142 + Pembrolizumab

SUMMARY:
A Phase 1/2 multicenter, dose determining, open-label study of ADXS31-142 monotherapy and a combination of ADXS31-142 and pembrolizumab (MK-3475) in participants with metastatic castration-resistant prostate cancer. Part A will be dose-determining part of ADXS31-142 monotherapy. Part B will be dose-determining part of ADXS31-142 and pembrolizumab (MK-3475) in combination. Part B expansion will treat additional participants with the recommended dose from Part B.

DETAILED DESCRIPTION:
Part A of the study will be an open-label, Phase 1, multicenter, non-randomized, dose-determining trial of ADXS31-142 monotherapy in participants with mCRPC. The dose determining phase is intended to select a recommended Phase 2 dose (RP2D) for Part B.

Part B of the study will be an open-label, Phase 1-2, multicenter, non-randomized dose-determining trial of ADXS31-142 in combination with pembrolizumab (MK-3475) in participants with mCRPC. Part B will consist of a dose-determination phase followed by an expansion cohort phase. The dose-determining phase is intended to select an RP2D for the combination.

Dose escalation/de-escalation for this study will be explored by applying the modified toxicity probability interval design.

ELIGIBILITY:
Inclusion Criteria:

1. Have progressive mCRPC, on androgen deprivation therapy, based on at least one of the following criteria:

   1. Prostate-specific antigen (PSA) progression, defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval with a minimum PSA of 2 ng/mL.
   2. Progression of bi-dimensionally measurable soft tissue (nodal metastasis) assessed within 1 month prior to registration by computed tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen and pelvis.
   3. Progression of bone disease (evaluable disease) (new bone lesion[s]) by bone scan.
2. Has discontinued antiandrogens (bicalutamide, nilutamide) >6 weeks and enzalutamide >4 weeks prior to Day 1 of trial treatment
3. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.

Exclusion Criteria:

1. Received more than 3 prior systemic treatment regimens with chemotherapy, hormonal, or immunotherapy in the metastatic setting or received more than 1 prior chemotherapeutic regimen in the metastatic setting
2. Has a diagnosis of immunodeficiency or is receiving any systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Day 1 of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., Grade ≤1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., Grade ≤1 or at baseline) from adverse events due to a previously administered agent.
5. Has received prior therapy with an anti-programmed cell death protein-1 (PD-1), anti-programmed death-ligand-1 (PD-L1), or anti-Programmed death-ligand-2 (PD-L2) agent or if the participant has previously participated in a Merck MK-3475 clinical trial.
6. Has a contraindication to administration of ampicillin or trimethoprim/ sulfamethoxazole.
7. Has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants, and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device and/or implant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Recruiting, San Francisco, California
  - University of Colorado Health Sciences Center (UCHSC), Aurora, Colorado
  - Recruiting, Rockville, Maryland
  - Recruiting, Towson, Maryland
  - New Brunswick, New Jersey
  - Recrutiing, Philadelphia, Pennsylvania
  - Site, Philadelphia, Pennsylvania
  - Recruiting, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stein MN, Fong L, Tutrone R, Mega A, Lam ET, Parsi M, Vangala S, Gutierrez AA, Haas NB. ADXS31142 Immunotherapy +/- Pembrolizumab Treatment for Metastatic Castration-Resistant Prostate Cancer: Open-Label Phase I/II KEYNOTE-046 Study. Oncologist. 2022 Jun 8;27(6):453-461. doi: 10.1093/oncolo/oyac048. PMID 35373299
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9177110/

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: ADXS31-142 1x10^9 CFU: Participants received ADXS31-142 1 × 10^9 CFU intravenously (IV) every 3 weeks (Q3W) in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 5×10^9 CFU: Participants received ADXS31-142 5 × 10^9 CFU intravenously (IV) every 3 weeks (Q3W) in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 1×10^10 CFU: Participants received ADXS31-142 1 × 10^10 CFU intravenously (IV) every 3 weeks (Q3W) in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part B: ADXS31-142 1×10^9 CFU + Pembrolizumab: Participants received ADXS31-142 1 × 10^9 CFU IV Q3W (in a 12-week cycle) in combination with 200 mg pembrolizumab IV Q3W for three times, with a fourth pembrolizumab dose 3 weeks later (in 12 week-cycles) for up to 24 months or until disease progression or discontinuation.
Period: Overall Study
Arm/Group | Part A: ADXS31-142 1x10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 1×10^9 CFU + Pembrolizumab
Started | 10 | 1 | 2 | 37
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 1 | 2 | 37
Not completed — Progressive disease | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 15
Not completed — Death | 5 | 1 | 1 | 16
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: The All Treated Population included all participants who received at least one dose of ADXS31-142 or pembrolizumab.
Groups:
- Part A: ADXS31-142 1×10^9 CFU: Participants received ADXS31-142 1 × 10^9 CFU intravenously (IV) every 3 weeks (Q3W) in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part B: ADXS31-142 + Pembrolizumab: Participants received ADXS31-142 1 × 10^9 CFU IV Q3W (in a 12-week cycle) in combination with 200 mg pembrolizumab IV Q3W for three times, with a fourth pembrolizumab dose 3 weeks later (in 12 week-cycles) for up to 24 months or until disease progression or discontinuation.
- Total: Total of all reporting groups
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab | Total
Number analyzed (Participants) | 10 | 1 | 2 | 37 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 0 | 11 | 14
  >=65 years | 7 | 1 | 2 | 26 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 1 | 2 | 37 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 1 | 2 | 36 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 7 | 7
  White | 9 | 1 | 2 | 30 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Adverse events with onset dates on or after the first dose of study medication and within 30 days following the last dose of study medication were considered "treatment emergent".
Time Frame: From first dose up to 30 days after last dose (maximum duration: 108 weeks)
Population: The All Treated Population included all participants who received at least one dose of ADXS31-142 or pembrolizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: ADXS31-142 1×10^9 CFU: Participants received ADXS31-142 1 × 10^9 CFU, IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 5×10^9 CFU: Participants received ADXS31-142 5×10^9 CFU, IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- ADXS31-142 1×10^10 CFU: Participants received ADXS31-142 1×10^10 CFU, IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
Number analyzed (Participants) | 10 | 1 | 2 | 37
Participants | 10 | 1 | 2 | 37

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 was defined as the number of participants with objective evidence of radiologic complete response (CR: disappearance of all target lesions) and partial response (PR: at least a 30% decrease in the sum of the longest diameters of target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions) as determined from investigator response assessments. Disease Control Rates are based upon confirmed events only.
Time Frame: From screening until progression or death (maximum duration: 104 weeks)
Population: The ORR Evaluable Population included all participants who received at least one dose of ADXS31-142 or pembrolizumab and who had at least one post-baseline radiologic tumor response assessment (CR, PR, stable disease [SD], or progressive disease [PD]) with evaluable results.
Measure: Number; unit: participants
Groups:
- Part A: ADXS31-142 1×10^9 CFU: Participants received ADXS31-142 1 × 10^9 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 5×10^9 CFU: Participants received ADXS31-142 5 × 10^9 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 1×10^10 CFU: Participants received ADXS31-142 1 × 10^10 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
Number analyzed (Participants) | 7 | 1 | 0 | 29
participants | 0 | 0 |  | 0

3. Secondary Outcome: Objective Response Rate According to Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: The ORR according to irRECIST was defined as the number of participants with objective evidence of radiologic immune-related CR (irCR: Disappearance of all target lesions) and immune-related PR (irPR: At least 30% decrease in tumor burden compared with baseline) as determined from investigator response assessments.
Time Frame: From screening until progression or death (maximum duration: 104 weeks)
Population: Participants in the ORR Evaluable Population were analyzed. The ORR Evaluable Population included all participants who received at least one dose of ADXS31-142 or pembrolizumab and who had at least one post-baseline radiologic tumor response assessment (CR, PR, stable disease [SD], or progressive disease [PD]) with evaluable results.
Measure: Number; unit: participants
Groups:
- Part A: ADXS31-142 1×10^9 CFU: Participants received ADXS31-142 1×10^9 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
- Part A: ADXS31-142 5×10^9 CFU: Participants received ADXS31-142 5×10^9 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
Number analyzed (Participants) | 7 | 1 | 0 | 28
participants | 0 | 0 |  | 0

4. Secondary Outcome: Progression-free Survival, Assessed by RECIST Version 1.1
Description: Progression-free survival (PFS) was defined as the time from randomization until objective tumor progression based on response evaluation criteria in solid tumors (RECIST) version 1.1 or death. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions. Participants who had not experienced disease progression or who were still alive at the time of evaluation were censored for the analysis. The PFS was estimated using Kaplan-Meier method.
Time Frame: From screening until progression or death (maximum duration: 104 weeks)
Population: All treated patients population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part A: ADXS31-142 1×10^10 CFU: Participants received ADXS31-142 1×10^10 CFU, IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
Number analyzed (Participants) | 10 | 1 | 2 | 37
Months | 2.2 [0.8 to NA] — lack of events due to censoring | NA [NA to NA] — lack of events due to censoring | NA [NA to NA] — lack of events due to censoring | 5.3 [2.1 to 7.9]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of start of study treatment until death due to any cause. Any participant not died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. The OS was estimated using Kaplan-Meier method.
Time Frame: From screening until progression or death (maximum duration: 104 weeks)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
Number analyzed (Participants) | 10 | 1 | 2 | 37
Months | 7.8 [1.3 to NA] — Sample size is too small. Lack of events due to censoring | 18.5 [NA to NA] — Sample size too small | 7.8 [NA to NA] — Sample size is too small. Lack of events due to censoring | 33.7 [15.4 to NA] — The upper 95% CI cannot be calculated due to insufficient number of events in the tested time frame

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose (maximum duration: 108 weeks)
Description: The All Treated Population included all participants who received at least one dose of ADXS31-142 or pembrolizumab.
Groups:
- Part A: ADXS31-142 1×10^10 CFU: Participants received ADXS31-142 1×10^10 CFU IV Q3W in a 12-week cycle for up to 24 months or until disease progression or discontinuation.
Arm/Group | Part A: ADXS31-142 1×10^9 CFU | Part A: ADXS31-142 5×10^9 CFU | Part A: ADXS31-142 1×10^10 CFU | Part B: ADXS31-142 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/10 | 1/1 | 1/2 | 16/37
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/1 | 1/2 | 22/37
Other Adverse Events (participants affected / at risk) | 10/10 | 1/1 | 2/2 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ADXS31-142 1×10^9 CFU (N=10) | Part A: ADXS31-142 5×10^9 CFU (N=1) | Part A: ADXS31-142 1×10^10 CFU (N=2) | Part B: ADXS31-142 + Pembrolizumab (N=37)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 3 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cerebral ischemia (Nervous system disorders) | 0 | 0 | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone Neoplasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Iiird Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ADXS31-142 1×10^9 CFU (N=10) | Part A: ADXS31-142 5×10^9 CFU (N=1) | Part A: ADXS31-142 1×10^10 CFU (N=2) | Part B: ADXS31-142 + Pembrolizumab (N=37)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 4
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 9
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 4
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 5
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 19
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 9
Asthenia (General disorders) | 2 | 1 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 7 | 1 | 2 | 34
Face oedema (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 4 | 1 | 0 | 14
Gait disturbance (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 0 | 9
Pain (General disorders) | 1 | 0 | 0 | 6
Pyrexia (General disorders) | 7 | 1 | 1 | 21
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 6
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 8
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 4
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2 | 8
Hypotension (Vascular disorders) | 3 | 1 | 2 | 7
Eye Pain (Eye disorders) | 0 | 1 | 0 | 0
Eyelid Ptosis (Eye disorders) | 0 | 1 | 0 | 0
Orbital Oedema (Eye disorders) | 0 | 1 | 0 | 0
Anal Sphincter Atony (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Temperature Intolerance (General disorders) | 0 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Radiation Associated Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases To Bone Marrow (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Metastases To Nasal Sinuses (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall seek the Sponsor's written approval for study results publication which shall not be unreasonably withheld. Such publication by Institution and/or Investigator may be no earlier than after a cooperative publication has been published with Sponsor or 1 year from date of completion or termination of the Study & only after review and comment by Sponsor. Institution agrees to provide Sponsor a copy of proposed publication at least 60 days prior to submission to a publisher.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02325557/Prot_SAP_000.pdf